CLINICAL TRIAL: NCT07121751
Title: Optimal Stimulation of Hypo-responders Undergoing IVF: a Prospective, Randomized, Controlled Trial
Brief Title: Optimal Stimulation of Hypo-responders Undergoing in Vitro Fertilization (IVF)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dunamenti REK Istenhegyi IVF Center (Other)
Collaborators: Dunamenti REK Gyor Clinic (Unknown); Dunamenti REK Pannon Clinic (Unknown); University of Szeged, Hungary (Unknown)
Responsible Party: Principal Investigator, Peter Kovacs MD, medical director Dunamenti REK Istenhegyi IVF Center, Dunamenti REK Istenhegyi IVF Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNGYK/22108-7/2025
Record Dates: First submitted 2025-07-25; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hypo-responder; Infertility (IVF Patients); OVARIAN STIMULATION
Keywords: ovarian stimulation; in vitro fertilization; hypo-responder; gonadotropin; luteinizing hormone
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): In this arm the hypo-responder patient will undergo stimulation using the same gonadotropin dose as in her previous treatment.
  Treatment steps:
  1. Stimulation using the same recombinant FSH dose as in her prevoius cycle is started on day 2 or 3 of the menstrual cycle and is continued for 5 days. On day 6 the patient is seen for US and bloodwork. If indicated the dose can be increased by max. 75 IU every 2 days to a maximum of 300 IU/day.
  2. GnRH antagonist is started at follicle size 12-14 m.
  3. Trigger is administered once the largest follicle gets >17 mm. Retrieval is scheduled 36 hrs later. IVF or ICSI fertilization. Luteal support from day past retrieval.
  4. Transfer of 1-2 embryos on day 3 or 5.
  5. Pregnancy test 12 days after ET.
  Interventions: Drug: unchanged dose
- Additional LH group (Pergoveris, Merck) (Active Comparator): In this arm the hypo-responder patient will undergo stimulation using the same gonadotropin dose as in her previous treatment but in the form of rec FSH and recLH 2:1 ratio (e.g.: if 150 IU rec FSH was used then 150 IU recFSH and recLH (2:1 ratio).
  Treatment steps:
  1. Stimulation using the same dose as in her previuos cycle but in the form of recombinant FSH and recombinant LH 2:1 ratio is started on day 2 or 3 of the menstrual cycle and is continued for 5 days. On day 6 the patient is seen for US and bloodwork. If indicated the dose can be increased by max. 75 IU every 2 days to a maximum of 300 IU/day.
  2. GnRH antagonist is started at follicle size 12-14 m.
  3. Trigger is administered once the largest follicle gets >17 mm. Retrieval is scheduled 36 hrs later. IVF or ICSI fertilization. Luteal support from day past retrieval.
  4. Transfer of 1-2 embryos on day 3 or 5.
  5. Pregnancy test 12 days after ET.
  Interventions: Drug: use of combination of recombinant FSH and recombinant LH
- higher dose FSH group (follitropin alpha (Gonal-F, Ovaleap) or follitropin delta (Rekovelle) (Active Comparator): In this arm the hypo-responder patient will undergo stimulation using recombinant FSH but with a dose increase of 75 IU/day compared to the gonadotropin dose used in her previous treatment (e.g.: if 150 IU/d rec FSH was used then 225 IU/d will be used).
  Treatment steps:
  1. Stimulation using an additional 75 IU recombinant FSH per day compared to her previous treatment is started on day 2 or 3 of the menstrual cycle and is continued for 5 days. On day 6 the patient is seen for US and bloodwork. If indicated the dose can be increased by max. 75 IU every 2 days to a maximum of 300 IU/day.
  2. GnRH antagonist is started at follicle size 12-14 m.
  3. Trigger is administered once the largest follicle gets >17 mm. Retrieval is scheduled 36 hrs later. IVF or ICSI fertilization. Luteal support from day past retrieval.
  4. Transfer of 1-2 embryos on day 3 or 5.
  5. Pregnancy test 12 days after ET.
  Interventions: Drug: higher dose recFSH

INTERVENTIONS:
Drug: use of combination of recombinant FSH and recombinant LH — in this arm the patients will use the combination of recFSH:recLH in the same dose as in her prior cycle
  Arms: Additional LH group (Pergoveris, Merck)
Drug: higher dose recFSH — in this arm the patient will use an additional 75 IU/day recFSH compared to her previous drug dose
  Arms: higher dose FSH group (follitropin alpha (Gonal-F, Ovaleap) or follitropin delta (Rekovelle)
Drug: unchanged dose — in this groups the patient will receive the same recFSH dose as in her prior cycle
  Arms: Control group

SUMMARY:
Stimulation is a key step of in vitro fertilization (IVF). Typically, injectable gonadotropins are used for stimulation, and their dose is individually determined to avoid hypo- as well as hyper-response. Despite the individualization some patients respond with a lower-than-expected number of oocytes. If the low response is unexpected based on the baseline parameters or if an unusually high dose of gonadotropins is needed to achieve a proper response we talk about "hypo-response". In such cases if the first treatment fails and a repeat attempt is planned typically even more gonadotropins, the combination of luteinizing hormone (LH) with follicle stimulating hormone (FSH) or the use of the more potent recombinant preparations are considered. The benefits of these approaches however have not been studied properly in hypo-responders. The studies have used various criteria to identify hypo-responders, have used various gonadotropin doses and have evaluated different outcome parameters. Live birth was only studied in one trial.

It is also known that in a different cycle the same patient is likely to have a slightly different response to the same type and dose of drugs. Therefore, the question arises whether a hypo-responder in one treatment is expected to have hypo-response again if the treatment is similarly carried out in a different cycle. Do we need to change/ increase the gonadotropin dose if based on age and ovarian reserve otherwise we would expect a normal response? Furthermore, if we consider a change should we increase the dose of FSH or should we combine it with LH?

Therefore the aim of this randomized controlled trial is compare an unchanged medication regimen to increased dose of FSH vs the combination of FSH and LH in hypo-responder patients identified based on POSEIDON (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number) criteria (Gr 1 and 2: retrieval of 9 or fewer oocytes in patients with an anti-Müllerian hormone (AMH) level ≥ 1.2 ng/ml or antral follicle count (AFC) ≥ 5 and age <35 years [Group (Gr) 1] or ≥35 years [Gr2]). Hypo-responder patients will be randomized to:

1. Same gonadotropin dose as in previous treatment (recombinant(r) FSH) ['control group']
2. The same dose as in the previous cycle but in the form of FSH + LH combination (rFSH:rLH 2:1 ratio) ['additional LH group']
3. A dose increase of 75 international unit (IU) compared to the dose in the previous treatment. ['higher dose FSH group'] The primary outcome parameter to study is live clinical pregnancy. In addition, baseline demographic, stimulation and further clinical outcomes (pregnancy rate, miscarriage rate, live birth rate) will be compared.

DETAILED DESCRIPTION:
The key step of an IVF treatment is controlled ovarian stimulation. The aim of stimulation is to recruit an optimal number of oocytes. The outcome of the fresh cycle improves if the collected oocyte number increases up to 10-15 oocytes. Cumulative success however keeps on rising even over 20 oocytes.

In most of the IVF cycles injectable gonadotropins are used to induce multi-follicular development. The type and dose of the gonadotropins are individually determined based on age, ovarian reserve markers, weight and previous response to treatment. Based on these parameters patients are grouped as expected low-, normal- or high-responders.

Despite a seemingly adequate stimulation regimen some patients respond with fewer than the expected number of follicles/ oocytes. Such patients are called hypo-responders. According to the POSEIDON classification these patients belong to POSEIDON groups 1 and 2 (Gr 1 and 2: retrieval of 9 or fewer oocytes in patients with an anti-Müllerian hormone (AMH) level ≥ 1.2 ng/ml or antral follicle count (AFC) ≥ 5 and age <35 years [Gr1] or ≥35 years [Gr2]). Other definitions to identify hypo-responders are: 1) use of >2500 IU gonadotropins during stimulation, 2) lack of follicle growth during stimulation, 3) lack of estradiol rise during stimulation. In these cases, we expect a proper response, but it either does not happen, or we need to administer high doses of gonadotropins to achieve the desired result. The exact cause of this phenomenon is not known but receptor polymorphism is one mechanism that could interfere with appropriate signal transduction. Another hypothesis is that these patients are less sensitive to LH and despite adequate serum LH levels they suffer from a reduced LH effect.

If a hypo-responder patient needs to undergo a second treatment, usually either the gonadotropin dose is increased from the onset of the stimulation, or the FSH preparation is combined with LH, or the more potent recombinant preparations are favored. LH could play a dual role; it increases androgen synthesis in the theca cells which in turn increases the FSH sensitivity and aromatase activity of the granulosa cells. In addition, mid-size follicles express LH receptors and therefore LH can directly support their development.

According to one meta-analysis, if treatment outcome is compared with rFSH vs rFSH+rLH in the general, non-selected population then with rFSH more oocytes can be collected while the rFSH+rLH combination results in more pregnancies. Another meta-analysis focusing on poor responders found more oocytes and higher clinical pregnancy rates after rFSH+rLH treatment but no difference in the live birth rates.

However, only a few properly designed studies have compared the various treatment strategies among hypo-responders. Lisi et al. have supplemented with rLH from day 7 onwards the second stimulation of those patients who required >2500 IU gonadotropin in their first attempt. Clinical pregnancy rate was higher in the rLH supplemented cycles. Based on these findings the authors designed a quasi-randomized trial during which every 3rd patient was given rLH supplementation from day 7 onwards. Among those who eventually needed >2500 IU gonadotropin those who were supplemented with rLH had higher implantation rates. There were however only 8 such cases. Ferraretti et al., have studied patients who had stagnation of follicle growth and estradiol production between days 7-10 of their treatment. The participants either received a higher FSH dose or received the combination or rFSH+rLH or the combination of rFSH + human menopausal gonadotropins (hMG). With rFSH alone the number of oocytes, the estradiol level and the clinical pregnancy rate were lower, but the live birth rate did not differ among the three groups. De Placido et al., in a study with a similar design to Ferraretti et al. found more oocytes in the increased rFSH dose arm but clinical outcome remained comparable in the three arms. In a study by Ruolvo et al., among women who needed >3000 IU gonadotropins previously the combination of rFSH with rLH resulted in more pregnancies. Finally, Yilmaz et al. reported improved implantation and pregnancy rates in hypo-responders with the combination of rFSH+rLH. Conforti et al., in a meta-analysis of trials in hypo-responders found that with rFSH+rLH an additional 2 oocytes can be collected and the live birth rate increases.

It is also known from daily practice that the same patient can respond differently to the same medication type and dose in a different cycle. Folliculogenesis is a long process lasting 3-6 months and most of this process is independent of gonadotropins. Those follicles that enter the final 2-3 weeks of this process become responsive to FSH and LH. The size of these groups of follicles varies from cycle to cycle. Therefore, the question arises whether a hypo-responder in one treatment is expected to have a similar hypo-response if the treatment is carried out without alterations. Do the providers need to change/ increase the gonadotropin dose if otherwise based on age and ovarian reserve one would expect a normal response? Furthermore, if adjustments are considered should the dose of FSH be increased or should a mixture with LH be used? In order to try to answer these question the investigators plan to perform a randomized controlled trial.

The aim of this randomized controlled trial is compare unchanged medication protocol to increased dose of FSH vs the combination of FSH and LH in hypo-responder patients identified based on POSEIDON criteria.

Inclusion criteria:

* indication for IVF- intracytoplasmic sperm injection (ICSI)
* age 18-40 years
* <9 oocytes in a previous IVF cycle and having an AMH ≥1.2 ng/ml and/or AFC ≥5 (POSEIDON 1,2)
* The use of ≤225 IU FSH (either rFSH alone or the combination of rFSH+human Menopausal Gonadotropin (hMG)) in the previous cycle
* regular 24-35 day cycles
* Intact uterine cavity
* motile sperm from ejaculate or testicular biopsy Exclusion criteria
* not meeting the inclusion criteria
* the use of rFSH:rLH (2:1 ratio) in the previous cycle
* the use of clomiphene citrate or aromatase inhibitor in the previous cycle
* >225 IU gonadotropin in the previous cycle
* >3 failed previous treatments
* patient with recurrent miscarriages
* presence of a hydrosalpinx
* positive human immunodeficiency virus (HIV) or hepatitis screening test
* planned preimplantation genetic testing of the embryos
* planned elective cryopreservation
* lack of consent Randomization: An online randomization list will be accessible from all participating centers by the local primary investigator using a personal link (www.randomizer.org). The other participating providers will receive the assignment from the local principle investigator (PI) once the patient has signed the consent form.

Sample size: Considering the pilot nature of the study the investigators plan to enroll 50 patients per treatment arm, 150 in total. If one treatment proves to be superior to the others, then the results could serve as the basis for a larger properly powered study.

Study sites: 4 IVF centers will participate: Dunamenti REK Istenhegyi IVF Center, Dunamenti REK Gyor IVF Center, Dunamenti REK Tapolca IVF Center, Reproductive Medicine Institute University of Szeged.

Outcome parameters:

* primary outcome: live clinical pregnancy at week 10-12 of gestation
* secondary outcomes: pregnancy rate, clinical pregnancy (intrauterine gestational sac), live birth rate (birth a live newborn after week 24 of gestation), miscarriage rate, birth weight, week of delivery

Definitions:

* Biochemical pregnancy: hCG>10 IU/l
* Clinical pregnancy: intrauterine gestational sac
* Ongoing pregnancy: embryo with heartbeat at week 10-12
* Early miscarriage: pregnancy loss prior to week 12
* Late miscarriage: pregnancy loss week 12-24
* Live birth: delivery after 24 weeks gestation
* Preterm delivery: delivery prior to week 37 gestation
* Very preterm delivery: delivery before week 32 gestation
* Low birth weight: < 2500 g
* Very low birth weight: < 1500 g

Treatment arms:

1. Same gonadotropin dose as in previous treatment (recombinant(r) FSH) ['control group']
2. The same dose as in the previous cycle but in the form of FSH + LH combination (rFSH:rLH 2:1 ratio) ['additional LH group']
3. A dose increase of 75 IU compared to the dose in the previous treatment. ['higher dose FSH group']

Treatment plan:

1. The patient meeting the inclusion or exclusion criteria is seen for an ultrasound during the cycle preceding the IVF treatment and is randomized according to the online list after consent has been given.
2. Stimulation is started on day 2 or 3 of the menstrual cycle and is continued for 5 days. On day 6 the patient is seen for transvaginal ultrasound to assess the size and number of follicles and undergoes blood test for estradiol and LH. If the provider decides to increase the dose of the medication, then it can be increased by max. 75 IU every 2 days to a maximum of 300 IU/day.
3. Once the largest follicles reach 12-14 mm in diameter 0.25 mg cetrorelix (Gonadotropin-releasing hormone (GnRH) antagonist) is started.
4. At the time of the last follicle scan serum estradiol, progesterone and LH levels are measured again.
5. Once the largest follicle reaches >17 mm in diameter the trigger injection (recombinant human chorionic gonadotropin (rHCG) or the combination of rHCG + GnRH agonist) is administered or if the provider considers the risk of ovarian hyperstimulation syndrome (OHSS) to be high pure GnRH agonist trigger (with elective cryopreservation) can be administered.
6. 35-36 hours after the trigger transvaginal oocyte retrieval is performed. Fertilization by IVF or ICSI depending on the semen parameters and patient history.
7. Vaginal progesterone supplementation from the day after the retrieval.
8. 3-5 days after the retrieval 1-2 embryos/blastocysts are transferred transcervically. Surplus good morphology embryos are cryopreserved using vitrification.
9. 12-14 days after the transfer serum beta HCG test to confirm pregnancy.
10. If the test is positive in another 3+/-0.5 weeks ultrasound to confirm intrauterine implantation.
11. Second ultrasound to confirm live ongoing pregnancy around week 10.
12. Luteal support up to week 8-9 of gestation.
13. Follow up until delivery to collect perinatal outcome parameters.
14. If the first transfer fails but frozen embryos are available frozen embryo transfer (FET) can be planned.

Parameters to be collected:

* age
* number of previous embryo transfers
* indication for IVF
* body mass index
* smoking history
* day 6 estradiol + LH levels
* estradiol, LH, progesterone at last scan
* endometrial thickness at last scan
* number of oocytes
* number of mature oocytes
* method of fertilization
* number of fertilized oocytes
* number of embryos
* number of embryos transferred
* number of embryos cryopreserved
* embryo quality (Gardner score in case of blastocysts)
* result of the initial hCG
* clinical pregnancy
* live clinical pregnancy
* miscarriage
* live birth
* week of delivery
* birth weight
* adverse events: 1) elevated progesterone prior to retrieval (>1.5 ng/ml), 2) elective cryopreservation for OHSS, 3) OHSS, 4) other (complications during retrieval)

Statistical methods:

Statistical analysis: Baseline demographic, IVF treatment related, and clinical outcomes will be compared in the three different stimulation protocol groups. Continuous variables will be shown as mean +/- standard deviation (SD), while categorical variable as number and percent. ANOVA and Mann-Whitney U test will be used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* indication for IVF-ICSI
* age 18-40 years
* <9 oocytes in a previous IVF cycle and having an AMH ≥1.2 ng/ml and/or AFC ≥5 (POSEIDON 1,2)
* The use of ≤225 IU FSH (either rFSH alone or the combination of rFSH+hMG) in the previous cycle
* regular 24-35 day cycles
* Intact uterine cavity
* motile sperm from ejaculate or testicular biopsy

Exclusion Criteria:

* not meeting the inclusion criteria
* the use of rFSH:rLH (2:1 ratio) in the previous cycle
* the use of clomiphene citrate or aromatase inhibitor in the previous cycle
* >225 IU gonadotropin in the previous cycle
* >3 failed previous treatments
* patient with recurrent miscarriages
* presence of a hydrosalpinx
* positive HIV or hepatitis screening test
* planned preimplantation genetic testing of the embryos
* planned elective cryopreservation
* lack of consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
live clinical pregnancy | up to 3 months after the embryo transfer; starting with the first patient who has a positive pregnancy test after transfer and up to 3 months after the completion of the study (last transfer with positive result)
  intrauterine gestational sac with an embryo with heartbeat at week 10-12

SECONDARY OUTCOMES:
live birth | from up to 9 month after the embryo transfer; starting with the first patient who has a positive pregnancy test after the embryo transfer and up to 8 months after the completion of the study (last transfer with positive result)
  Live birth: delivery after 24 weeks gestation

OTHER OUTCOMES:
Biochemical pregnancy | starting 2 weeks after the first transfer and up to 2 weeks after the last embryo transfer
  hCG>10 IU/l 12-14 days after embryo transfer
Early miscarriage | starting 4 weeks after the first positive pregnancy test and up to 12 weeks after the last positive pregnancy test after the completion of the study (last transfer with positive result)
  loss of a clinical pregnancy prior to week 12
late miscarriage | starting 12 weeks plus 1 day after the first positive pregnancy test and up to 24 weeks after the last positive pregnancy test after the completion of the study (last transfer with positive result)
  pregnancy loss week 12-24
Live birth | starting 24 weeks plus 1 day after the first positive pregnancy test and up to 8 months after the last positive pregnancy test after the completion of the study (last transfer with positive result)
  delivery after 24 weeks gestation
preterm delivery | starting 24 weeks plus 1 day after the first positive pregnancy test and up to 7 months after the last positive pregnancy test after the completion of the study (last transfer with positive result)
  delivery prior to week 37 gestation
very preterm delivery | starting 24 weeks plus 1 day after the first positive pregnancy test and up to 5.5 months after the last positive pregnancy test after the completion of the study (last transfer with positive result)
  delivery before week 32 gestation
low birth weight | starting 24 weeks plus 1 day after the first positive pregnancy test and up to 8 months after the last positive pregnancy test after the completion of the study (last transfer with positive result)
  birth weight less than 2500 grams
very low birth weight | starting 24 weeks plus 1 day after the first positive pregnancy test and up to 8 months after the last positive pregnancy test after the completion of the study (last transfer with positive result)
  birth weight less than 1500 grams

CONTACTS AND LOCATIONS:
Locations (4):
- Hungary (4):
  - Dunamenti REK Istenhegyi IVF Center, Budapest
  - Dunamenti REK Gyor IVF Center, Győr
  - University of Szeged, Reproductive Medicine Institute, Szeged
  - Dunamenti REK Tapolca IVF Center, Tapolca

IPD SHARING:
Plan to Share IPD: Undecided
Patient data will be shared upon reasonable request.

REFERENCES:
- [Background] Yazici Yilmaz F, Gorkemli H, Colakoglu MC, Aktan M, Gezginc K. The evaluation of recombinant LH supplementation in patients with suboptimal response to recombinant FSH undergoing IVF treatment with GnRH agonist down-regulation. Gynecol Endocrinol. 2015 Feb;31(2):141-4. doi: 10.3109/09513590.2014.965675. Epub 2014 Sep 19. PMID 25237892
- [Background] Ruvolo G, Bosco L, Pane A, Morici G, Cittadini E, Roccheri MC. Lower apoptosis rate in human cumulus cells after administration of recombinant luteinizing hormone to women undergoing ovarian stimulation for in vitro fertilization procedures. Fertil Steril. 2007 Mar;87(3):542-6. doi: 10.1016/j.fertnstert.2006.06.059. Epub 2006 Nov 27. PMID 17126339
- [Background] De Placido G, Alviggi C, Perino A, Strina I, Lisi F, Fasolino A, De Palo R, Ranieri A, Colacurci N, Mollo A; Italian Collaborative Group on Recombinant Human Luteinizing Hormone. Recombinant human LH supplementation versus recombinant human FSH (rFSH) step-up protocol during controlled ovarian stimulation in normogonadotrophic women with initial inadequate ovarian response to rFSH. A multicentre, prospective, randomized controlled trial. Hum Reprod. 2005 Feb;20(2):390-6. doi: 10.1093/humrep/deh625. Epub 2004 Dec 2. PMID 15576390
- [Background] Ferraretti AP, Gianaroli L, Magli MC, D'angelo A, Farfalli V, Montanaro N. Exogenous luteinizing hormone in controlled ovarian hyperstimulation for assisted reproduction techniques. Fertil Steril. 2004 Dec;82(6):1521-6. doi: 10.1016/j.fertnstert.2004.06.041. PMID 15589853
- [Background] Lisi F, Rinaldi L, Fishel S, Lisi R, Pepe GP, Picconeri MG, Campbell A. Use of recombinant LH in a group of unselected IVF patients. Reprod Biomed Online. 2002 Sep-Oct;5(2):104-8. doi: 10.1016/s1472-6483(10)61610-0. PMID 12419032
- [Background] Lisi F, Rinaldi L, Fishel S, Lisi R, Pepe G, Picconeri MG, Campbell A, Rowe P. Use of recombinant FSH and recombinant LH in multiple follicular stimulation for IVF: a preliminary study. Reprod Biomed Online. 2001;3(3):190-194. doi: 10.1016/s1472-6483(10)62034-2. PMID 12513853
- [Background] Lehert P, Kolibianakis EM, Venetis CA, Schertz J, Saunders H, Arriagada P, Copt S, Tarlatzis B. Recombinant human follicle-stimulating hormone (r-hFSH) plus recombinant luteinizing hormone versus r-hFSH alone for ovarian stimulation during assisted reproductive technology: systematic review and meta-analysis. Reprod Biol Endocrinol. 2014 Feb 20;12:17. doi: 10.1186/1477-7827-12-17. PMID 24555766
- [Background] Santi D, Casarini L, Alviggi C, Simoni M. Efficacy of Follicle-Stimulating Hormone (FSH) Alone, FSH + Luteinizing Hormone, Human Menopausal Gonadotropin or FSH + Human Chorionic Gonadotropin on Assisted Reproductive Technology Outcomes in the "Personalized" Medicine Era: A Meta-analysis. Front Endocrinol (Lausanne). 2017 Jun 1;8:114. doi: 10.3389/fendo.2017.00114. eCollection 2017. PMID 28620352
- [Background] Gougeon A. Regulation of ovarian follicular development in primates: facts and hypotheses. Endocr Rev. 1996 Apr;17(2):121-55. doi: 10.1210/edrv-17-2-121. No abstract available. PMID 8706629
- [Background] Conforti A, Esteves SC, Di Rella F, Strina I, De Rosa P, Fiorenza A, Zullo F, De Placido G, Alviggi C. The role of recombinant LH in women with hypo-response to controlled ovarian stimulation: a systematic review and meta-analysis. Reprod Biol Endocrinol. 2019 Feb 6;17(1):18. doi: 10.1186/s12958-019-0460-4. PMID 30728019
- [Background] Poseidon Group (Patient-Oriented Strategies Encompassing IndividualizeD Oocyte Number); Alviggi C, Andersen CY, Buehler K, Conforti A, De Placido G, Esteves SC, Fischer R, Galliano D, Polyzos NP, Sunkara SK, Ubaldi FM, Humaidan P. A new more detailed stratification of low responders to ovarian stimulation: from a poor ovarian response to a low prognosis concept. Fertil Steril. 2016 Jun;105(6):1452-3. doi: 10.1016/j.fertnstert.2016.02.005. Epub 2016 Feb 26. No abstract available. PMID 26921622
- [Background] Ovarian Stimulation TEGGO, Bosch E, Broer S, Griesinger G, Grynberg M, Humaidan P, Kolibianakis E, Kunicki M, La Marca A, Lainas G, Le Clef N, Massin N, Mastenbroek S, Polyzos N, Sunkara SK, Timeva T, Toyli M, Urbancsek J, Vermeulen N, Broekmans F. ESHRE guideline: ovarian stimulation for IVF/ICSIdagger. Hum Reprod Open. 2020 May 1;2020(2):hoaa009. doi: 10.1093/hropen/hoaa009. eCollection 2020. PMID 32395637
- [Background] Polyzos NP, Drakopoulos P, Parra J, Pellicer A, Santos-Ribeiro S, Tournaye H, Bosch E, Garcia-Velasco J. Cumulative live birth rates according to the number of oocytes retrieved after the first ovarian stimulation for in vitro fertilization/intracytoplasmic sperm injection: a multicenter multinational analysis including approximately 15,000 women. Fertil Steril. 2018 Sep;110(4):661-670.e1. doi: 10.1016/j.fertnstert.2018.04.039. PMID 30196963
- [Background] Fanton M, Cho JH, Baker VL, Loewke K. A higher number of oocytes retrieved is associated with an increase in fertilized oocytes, blastocysts, and cumulative live birth rates. Fertil Steril. 2023 May;119(5):762-769. doi: 10.1016/j.fertnstert.2023.01.001. Epub 2023 Jan 10. PMID 36634732